CLINICAL TRIAL: NCT01847586
Title: Enhancing Neuroplasticity and Frontal Lobe Function in Patients With Mild Alzheimer's Disease
Acronym: TMS-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tarek Rajji, Staff Psychiatrist and Clinician Researcher, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 215/2012
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Brain stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer's disease-rPAS (Experimental): The intervention procedure will done in this group is r-Paired Associative Stimulation. This involves the repetitive pairing of electrical stimulation of the median nerve with - 25 ms later - transcranial magnetic stimulation (TMS) of the contralateral DLPFC
  Interventions: Procedure: Paired Associative Stimulation
- Alzheimer's disease-rPAS-C (Placebo Comparator): The intervention procedure being done with this group is PAS-C. This is a control Paired Associative Stimulation paradigm in which TMS to the left DLPFC follows the electrical stimulation of the right median nerve by 100 ms, and, thus, does not result in contemporaneous occurrence of the two stimulations in the cortex and consequently no LTP.
  Interventions: Procedure: Paired Associative Stimulation-Control
- Control (Other): Controls will have a one time Paired Associative Stimulation-Control (PAS-C) paradigm intervention in which TMS to the left DLPFC follows the electrical stimulation of the right median nerve by 100 ms, and, thus, does not result in contemporaneous occurrence of the two stimulations in the cortex and consequently no LTP.
  Interventions: Procedure: Paired Associative Stimulation-Control

INTERVENTIONS:
Procedure: Paired Associative Stimulation — PAS simulates in humans the induction of long-term potentiation (LTP), a prototype of synaptic neuroplasticity. PAS involves the repetitive pairing of electrical stimulation of the median nerve with - 25 ms later - transcranial magnetic stimulation (TMS) of the contralateral DLPFC. As such, these two stimulations arrive simultaneously in the DLPFC and result in potentiation of TMS induced cortical evoked potential, analogous to in vitro LTP.
  Arms: Alzheimer's disease-rPAS
Procedure: Paired Associative Stimulation-Control — PAS-C is a control PAS paradigm in which TMS to the left DLPFC follows the electrical stimulation of the right median nerve by 100 ms, and, thus, does not result in contemporaneous occurrence of the two stimulations in the cortex and consequently no LTP.
  Arms: Alzheimer's disease-rPAS-C; Control

SUMMARY:
The purpose of this study is to determine if a novel brain stimulation approach using magnetic stimulation (Transcranial Magnetic Stimulation [TMS]) can improve memory and thinking processes in individuals with mild Alzheimer's disease (AD).

DETAILED DESCRIPTION:
In this study, the investigators aim at assessing and then enhancing neuroplasticity in the dorsolateral prefrontal cortex (DLPFC) and working memory - a key function of DLPFC - in patients with mild AD. The investigators will use a novel non-invasive brain stimulation approach, Paired Associative Stimulation (PAS). PAS simulates in humans the induction of long-term potentiation (LTP), a prototype of synaptic neuroplasticity. PAS involves the repetitive pairing of electrical stimulation of the median nerve with - 25 ms later - transcranial magnetic stimulation (TMS) of the contralateral DLPFC. As such, these two stimulations arrive simultaneously in the DLPFC and result in potentiation of TMS induced cortical evoked potential, analogous to in vitro LTP.

Specific Aim 1: To compare LTP in the DLPFC among patients with mild AD and healthy subjects.

Specific Aim 2: To assess the effect of a 2-week course of PAS (rPAS) as applied to the left DLPFC on LTP and performance on working memory in patients with mild AD in comparison with a 2-week course of PAS control condition (PAS-C, described below) (rPAS-C).

ELIGIBILITY:
Inclusion Criteria for patients:

* Age 65 or above
* Meet NINCDS-ADRDA and DSM-IV TR criteria for a current diagnosis of Alzheimer's Disease
* Stable does of acetylcholinesterase inhibitors for at least 3 months
* Willingness and ability to speak English
* Willingness and ability to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria for patients:

* Meets criteria for an Axis I diagnosis within the past 12 months other than Dementia of the Alzheimer type.
* Mini Mental Status Examination score of 16 or less as described above
* Meets diagnostic criteria for current alcohol or other drug dependence within 6 months of testing
* Electroconvulsive Therapy (ECT) within 6 months of testing.
* Left handedness.
* Incompetency to consent
* Any contraindication for TMS

Inclusion Criteria for healthy controls:

* Age 65 or above
* Willingness and ability to speak English
* Willingness and ability to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria for healthy controls:

* Meets criteria for an Axis I diagnosis other than simple phobias or adjustment disorder.
* Other neurological disorder affecting central nervous system.
* Psychotropic medication except for sedative /hypnotics at a stable dose for at least 4 weeks.
* Left handedness
* Any contraindication for TMS

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Paired Associated Stimulation induced Long-term potentiation as a measure of neuroplasticity in the dorsolateral prefrontal cortex | 14 days
  We are using a novel technique of TMS- EEG as developed by our group. Through this technique, not only motor evoked potential (MEP) but also cortical evoked activity (CEA) is recorded continuously while TMS is being delivered to the cortex. Thus, PAS-induced LTP could be indexed through the potentiation of not only MEP but also of CEA. TMS-EEG has been used by our group and others. Our group has used TMS-EEG in healthy individuals and patients with severe mental illness to study several neurophysiological phenomena in M1 and DLPFC such as cortical inhibition, gamma oscillations, and recently LTP.
  In summary, we propose to combine PAS with TMS-EEG to assess DLPFC neuroplasticity in patients with mild AD and then deliver a 2-week course of daily repetitive PAS (rPAS) to enhance DLPFC neuroplasticity and function as indexed by the N-back task. This will be measured to see if there are any changes after 1 day, 7 days and 14 days of the intervention procedure.

SECONDARY OUTCOMES:
N-back Task | pre-intervention (baseline) and then 1, 7, 14 days after intervention
  Working Memory Assessment: Participants will have their working memory assessed pre- and 1, 7, and 14 days post intervention using the N-back task. In the N-back task participants determine whether a stimulus is the same as that presented N trials back. One and 7 days post-intervention, the N-back task will be administered to assess the short- and long-term effect of rPAS on working memory as our preliminary data demonstrate a long-term enhancing effect of PAS on motor learning

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rajji, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar S, Zomorrodi R, Ghazala Z, Goodman MS, Blumberger DM, Daskalakis ZJ, Fischer CE, Mulsant BH, Pollock BG, Rajji TK. Effects of repetitive paired associative stimulation on brain plasticity and working memory in Alzheimer's disease: a pilot randomized double-blind-controlled trial. Int Psychogeriatr. 2023 Mar;35(3):143-155. doi: 10.1017/S1041610220003518. Epub 2020 Nov 16. PMID 33190659